CLINICAL TRIAL: NCT04850235
Title: Nab-paclitaxel Plus Cisplatin and Capecitabine as Neoadjuvant Chemotherapy Followed by Concurrent Chemoradiation for Locoregionally Advanced Nasopharyngeal Carcinoma: a Phase I Dose-escalation Study
Brief Title: Nab-paclitaxel Based TPX Neoadjuvant Chemotherapy for NPC Patients: a Dose-escalation Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-FXY-489
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TPX neoadjuvant chemotherapy +CCRT (Experimental): Patients receive neoadjuvant chemotherapy with Nab-PTX (150/175/200/225/250 mg/m2, D1) , cisplatin (75 mg/m2, D1) and capecitabine (1000 mg/m2, BID, D1-14) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100 mg/m2) concurrent every three weeks during radiotherapy (D1, D22, D43 of RT)
  Interventions: Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Nab paclitaxel — Nab paclitaxel plus cisplatin and capecitabine as neoadjuvant chemotherapy

SUMMARY:
Neoadjuvant chemotherapy followed by concurrent chemoradiation (CCRT) has been recommended in the treatment of locoregionally-advanced nasopharyngeal carcinoma (NPC), with docetaxel, cisplatin (DDP) and 5-fluorouracil (5-Fu) shown to be an effective regimen. Capecitabine is the precursor drug of 5-fluorouracil, and has been used in replace of 5-fluorouracil in NPC patients. Nab-paclitaxel (Nab-PTX) is a novel albumin-bound paclitaxel with a superior therapeutic index to docetaxel. We sought to find out the efficacy of Nab-PTX in three-drug triplet (Nab-PTX, DDP and capecitabine) and decide the best administration dose of Nab-PTX.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy followed by concurrent chemoradiation (CCRT) has been recommended in the treatment of locoregionally-advanced nasopharyngeal carcinoma (NPC), with docetaxel, cisplatin (DDP) and 5-fluorouracil (5-Fu) shown to be an effective regimen. Capecitabine is the precursor drug of 5-fluorouracil, and has been used in replace of 5-fluorouracil in NPC patients. Nab-paclitaxel (Nab-PTX) is a novel albumin-bound paclitaxel with a superior therapeutic index to docetaxel. It was developed to reduce toxicities associated with paclitaxel whilst maintaining or improving its chemotherapeutic effect. In vivo preclinical experiments have shown greater volume of distribution of nab-paclitaxel than paclitaxel, with similar half-life and clearance. The efficacy and optimal dose of Nab-PTX combined with DDP as doublet has been explored in metastatic NPC patients and locoregionally advanced patients, and it showed encouraging anti-tumor effects and manageable toxicities. However, what is the optimal dose of Nab-PTX and the efficacy of it in three-drug triplet (Nab-PTX, DDP and capecitabine) needs to be discovered. Therefore, this study aims to evaluate the efficacy and safety of Nab-PTX plus cisplatin and capecitabine neoadjuvant chemotherapy, followed by cisplatin-based concurrent chemoradiotherapy in the patients with locoregionally advanced nasopharyngeal carcinoma, to provide new evidence for the use of Nab-PTX in NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III.
2. Original clinical staged as III-IVa （according to the 8th AJCC edition).
3. No evidence of distant metastasis (M0).
4. Male and no pregnant female.
5. Satisfactory performance status: ECOG (Eastern Cooperative OncologyGroup) scale 0-1.
6. WBC ≥ 4×109 /L and PLT ≥100×109 /L and HGB ≥90 g/L.
7. With normal liver function test (ALT/AST ≤ 2.5×ULN, TBIL≤ 2.0×ULN).
8. With normal renal function test (Creatinine Clearance ≥ 60 ml/min ).

Exclusion Criteria:

1. Patients have evidence of relapse or distant metastasis.
2. Histologically confirmed keratinizing squamous cell carcinoma (WHO I).
3. Receiving radiotherapy or chemotherapy previously.
4. The presence of uncontrolled life-threatening illness.
5. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
6. Receiving other ways of anti-cancer therapy.
7. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | At the end of each cycle (each cycle is 21 days)
  If more than one-third of patients in a given cohort experienced a dose-limiting toxicity (DLT), enrollment will be stopped and the dose used in the previous cohort will be designated as the maximum tolerated dose
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | At the end of each cycle (each cycle is 21 days)
  Incidence rate of adverse events (AEs), evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria.

SECONDARY OUTCOMES:
Objective response rate | 3 months
  The proportion of patients whose tumors shrink to a certain size and maintain such size for a certain period of time, including patients with complete response (CR) and partial response (PR).
Disease control rate | 3 months
  The proportion of patients with response and stable disease (SD) after treatment, including patients with CR, PR and SD.
Overall survival | 2-year
  Overall survival is calculated from the date of enrollment to the date of the death from any cause or censored at the date of the last follow-up.
Progression-free survival | 2-year
  Progress-free survival is calculated from the date of enrollment to the date of the first progression at any site or death from any cause or censored at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yu-Chen, Luo MJ, Liu RP, Jin J, Deng SW, Tang LQ, Li XY, Liu LT, Luo DH, Sun R, Liu SL, Li JB, Liu Q, Wang P, Chen QY, Mai HQ, Guo SS. Phase I dose-escalation study of nab-paclitaxel combined with cisplatin and capecitabin as induction chemotherapy followed by concurrent chemoradiotherapy in patients with nasopharyngeal carcinoma. Radiother Oncol. 2024 Feb;191:110051. doi: 10.1016/j.radonc.2023.110051. Epub 2023 Dec 21. PMID 38135184